CLINICAL TRIAL: NCT03012100
Title: Double Blind, Parallel Groups, Controlled, Randomized Phase II Trial to Evaluate Vaccination With Folate Receptor Alpha Peptide Vaccine With GM-CSF as Vaccine Adjuvant Following Oral Cyclophosphamide Versus GM-CSF/Placebo to Prevent Recurrence in Patients With Triple Negative Breast Cancer
Brief Title: Multi-epitope Folate Receptor Alpha Peptide Vaccine, GM-CSF, and Cyclophosphamide in Treating Patients With Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RU011501I; NCI-2016-01878 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU011501I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-12-29; First posted 2017-01-06 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Bilateral Breast Carcinoma; Breast Inflammatory Carcinoma; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma; Unilateral Breast Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms; Unilateral Breast Neoplasms | interventions — Cyclophosphamide; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (FRalpha peptide vaccine, sargramostim) (Experimental): Patients receive cyclophosphamide PO BID on days 1-7 and 15-21 of cycle 1 only. Starting cycle 2, patients receive multi-epitope folate receptor alpha peptide vaccine with sargramostim ID on day 1. Treatment repeats every 28 days for cycles 2-7 and every 6 months for cycles 8-14 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Multi-epitope Folate Receptor Alpha Peptide Vaccine; Biological: Sargramostim
- Arm II (placebo, sargramostim) (Placebo Comparator): Patients receive cyclophosphamide as in Arm I. Starting cycle 2, patients receive placebo vaccine with sargramostim ID on day 1. Treatment repeats every 28 days for cycles 2-7 and every 6 months for cycles 8-14 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Biological: Sargramostim

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Multi-epitope Folate Receptor Alpha Peptide Vaccine — Given ID
  Other Names: FR Alpha Peptide Vaccine
  Arms: Arm I (FRalpha peptide vaccine, sargramostim)
Other: Placebo Administration — Given ID
  Arms: Arm II (placebo, sargramostim)
Biological: Sargramostim — Given ID
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This randomized phase II trial studies how well multi-epitope folate receptor alpha peptide vaccine, sargramostim (GM-CSF), and cyclophosphamide work to prevent the recurrence of stage 1-3 triple negative breast cancer. Vaccines made from a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving multi-epitope folate receptor alpha peptide vaccine, sargramostim (GM-CSF), and cyclophosphamide may work well together to prevent cancer recurrence after surgery and other standard treatments for triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that multi-epitope folate receptor alpha peptide vaccine (folate receptor [FR]alpha peptide vaccine) with sargramostim (GM-CSF) adjuvant will prolong the disease-free survival (DFS) compared to GM-CSF adjuvant treatment in patients with triple negative breast cancer.

SECONDARY OBJECTIVE:

I. To compare the safety and tolerability of metronomic cyclophosphamide followed by FRalpha peptide vaccine with GM-CSF versus GM-CSF alone.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine whether high level of antibody and cellular immune response toward the FRalpha measured at baseline is a prognostic factor for vaccine immune response and/or cancer relapse.

II. To determine whether the level of tumor expression of FRalpha at baseline is a prognosis factor for vaccine immune response and/or cancer relapse.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cyclophosphamide orally (PO) twice daily (BID) on days 1-7 and 15-21 of cycle 1 only. Starting cycle 2, patients receive multi-epitope folate receptor alpha peptide vaccine with sargramostim intradermally (ID) on day 1. Treatment repeats every 28 days for cycles 2-7 and every 6 months for cycles 8-14 in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cyclophosphamide as in Arm I. Starting cycle 2, patients receive placebo vaccine with sargramostim ID on day 1. Treatment repeats every 28 days for cycles 2-7 and every 6 months for cycles 8-14 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Female
* Resected unilateral or bilateral primary carcinoma of the breast without clinical evidence of metastatic disease (after neoadjuvant chemotherapy and/or adjuvant chemotherapy), negative for estrogen receptor (ER) and progesterone receptor (PR) (cut-off for positivity is > 10% positive tumor cells with nuclear staining), and negative for HER2 as defined by one of the four situations delineated below:

  * HER2 immunohistochemistry (IHC) expression of 0 or 1+ and in-situ hybridization non-amplified
  * HER2 IHC expression of 0 or 1+ and in-situ hybridization not done
  * HER2 IHC expression of 2+ and in-situ hybridization non-amplified
  * IHC not done and in-situ hybridization non-amplified
  * Note: central review is not required
  * Note: If biopsy and surgical specimens are discordant from each other with regard to ER, PR, and/or HER2 status, a patient will be allowed to enroll assuming at least one of the specimens meets the above criteria and no endocrine therapy use is planned going forward
* Completed planned breast CANCER surgeries, any radiation therapy, and any chemotherapy, whichever is last, >= 90 days but not >= 546 days prior to randomization

  * Note: Reconstructive and prophylactic surgeries are allowed after randomization (during study treatment)
* Patient had at least one of the following:

  * Biopsy or surgery-proven regional node involvement by cancer
  * T1c, T2, T3, or T4 disease (with inflammatory disease allowed) identified at the time of surgery or clinically identified prior to neoadjuvant chemotherapy
  * No complete response to neoadjuvant chemotherapy (those who did achieve complete response are still eligible if a pre-chemotherapy regional nodal biopsy identified cancer or if the pre-chemotherapy tumor measured > 1 cm)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 obtained =< 14 days prior to randomization
* Platelet count >= 75,000/uL obtained =< 14 days prior to randomization
* Aspartate transaminase (AST) =< 3 x upper limit of normal (ULN) obtained =< 14 days prior to randomization
* Creatinine =< 1.5 x ULN obtained =< 14 days prior to randomization
* Negative serum pregnancy test done =< 14 days prior to randomization, for women of childbearing potential only
* Provide informed written consent
* Willing to return to enrolling institution for follow-up
* Willing to provide tissue and blood samples for correlative research studies

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Clinical evidence of local recurrence or distant metastases; Note: New primary tumors are allowed, both contralaterally and ipsilaterally, but a prior breast cancer must have been more than 5 years beforehand
* Known hypersensitivity reaction to GM-CSF
* Active autoimmune disease that has required systemic treatment =< 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to randomization; Note: replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment; patients with vitiligo, Graves disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded; patients with Celiac disease controlled with diet modification are not excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

  * NOTE: Localized fungal or viral infections including of the skin, nails, mouth, and genital area are allowed
* History of other cancer < 5 years prior to consent (except non-melanoma skin cancer or carcinoma in situ of the uterine cervix) or current receipt of treatment another cancer (e.g., monoclonal antibody, small molecule pathway inhibitor)
* Treatment with systemic corticosteroid or immune-modulators =< 7 days prior to randomization
* Concurrent treatment with other experimental drugs or any other systemic anticancer therapy (due to unknown drug-vaccine potential interactions). Use of experimental or other targeted therapy > 3 months prior is allowed as long as it is not Her2-directed

  * NOTE: Aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), statins, and other medications commonly used to treat nononcologic, non-autoimmune conditions are allowed
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Prior or concurrent use of trastuzumab or other Her2-directed therapy
* Prior or concurrent use of a PD-1 or PD-L1 checkpoint inhibitor (including pembrolizumab) unless the use was >= 3 months prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Through study completion (average of 5 years)
  Will be estimated using the method of Kaplan-Meier. Will use the stratified log-rank tests.

SECONDARY OUTCOMES:
Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events 4.0 | Through study completion (average of 5 years)
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed by primary disease site to determine toxicity patterns. Will use the Cochran-Mantel Haenszel chi-squared test with study stratification factors. Will use logistic regression to test differences in proportions while controlling for the known covariates.
Overall survival | Through study completion (average of 5 years)
  Will be estimated using the method of Kaplan-Meier. Will use the stratified log-rank tests.
Vaccine induced folate receptor [FR]alpha-specific T cell responses defined as the proportion of patients with at least a 2-fold increase in the number of cells/plasma concentration | Through study completion (average of 5 years)
  Will be determined along with its corresponding 95% confidence interval.
FRalpha levels | Through study completion (average of 5 years)
  FRalpha levels at baseline will be examined as a prognostic factor in the vaccine immune response. A multivariable Cox proportional hazard model will be used to assess baseline FRalpha levels as a potential prognostic factor for immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Ruddy, Principal Investigator — Academic and Community Cancer Research United
Locations (12):
- United States (12):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin